CLINICAL TRIAL: NCT00487968
Title: Eltrombopag Pediatric Formulation Taste Testing in Healthy Adult Volunteers
Brief Title: Eltrombopag Taste Testing in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: TRA110087
Record Dates: First submitted 2007-06-15; First posted 2007-06-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2011-02

CONDITIONS: Healthy Subjects; Purpura, Thrombocytopenic, Idiopathic
Keywords: healthy adult volunteers; eltrombopag
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: eltrombopag

SUMMARY:
Based on a need for a pediatric formulation of eltrombopag for the treatment of pediatric thrombocytopenia, this study will help determine the best tasting pediatric formulation of eltrombopag. Healthy adult volunteers who are able to taste bitterness and who do not have a high sensitivity to bitterness will be enrolled. The subjects will evaluate different formulations and rate them based on the bitterness and effectiveness of sweetners. The outcome of this study will help support a decision for a new pediatric formulation of eltrombopag.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult based on a medical evaluation by a responsible physician
* male or female adult between 18 and 55 years old
* female subjects who are not pregnant or lactating
* females who are unable to have children must have documented medical verification
* females who are able to have children must have a negative pregnancy test
* capable of giving written informed consent

Exclusion criteria:

* subjects who are unable to taste bitterness or are extrememly sensitive to bitterness
* participated in a clinical trial within 30 days
* exposure to more than four new medicines within 12 months prior to the first day of dosing
* history of sensitivity to any of the study medications

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2007-05

PRIMARY OUTCOMES:
To establish a taste preference of eltrombopag in a pediatric formulation taken at initial dosing, 3hours, and 6 hours on Day 1 & 2. | at initial dosing, 3hours, and 6 hours on Day 1 & 2.

SECONDARY OUTCOMES:
Saftey will be monitored by: - vital signs and clinical labs will be taken at all visits | all visits
- physical exam and an echocardiogram (ECG) will be done at Day 1 & 2 | done at Day 1 & 2

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Overland Park, Kansas, United States